CLINICAL TRIAL: NCT03197714
Title: Phase Ib Clinical Trial of OPB-111077 in Patients With Relapsed or Refractory Acute Myeloid Leukaemia
Brief Title: Clinical Trial of OPB-111077 in Patients With Relapsed or Refractory Acute Myeloid Leukaemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry); Apices Soluciones S.L. (Industry); Vivia Biotech (Unknown)
Responsible Party: Principal Investigator, Joaquín Martínez López, MD, PhD, Head of Hematology Department, Hospital Universitario 12 de Octubre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDO-LMA-2016-01; 2016-004135-21 (EudraCT Number)
Record Dates: First submitted 2017-06-13; First posted 2017-06-23 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myeloid

STUDY DESIGN:
Intervention Model Description: Phase Ib, open-label, dose-escalation clinical trial to evaluate the best-tolerated doses in AML relapsed or refractory to chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- OPB-111077 (Experimental): Level 1: 200 mg daily Level 2: 250 mg daily
  Interventions: Drug: OPB-111077

INTERVENTIONS:
Drug: OPB-111077 — Two dose schemas will be employed:
  * Level 1: 200 mg daily
  * Level 2: 250 mg daily

SUMMARY:
Phase Ib, open-label, dose-escalation clinical trial to evaluate the best-tolerated doses in Acute Myeloid Leukaemia (AML) relapsed or refractory to chemotherapy.

This open-label, nonrandomized trial will comprise 2 stages. A dose escalation stage will characterize the safety, tolerability and maximum tolerated dose (MTD), of OPB-111077.

Subsequently, an expansion stage will further evaluate the safety and antitumor activity of OPB-111077 in AML relapsed or refractory to chemotherapy.

Enrollment to the expansion cohort will begin following determination of the MTD.

Approximately 6-12 patients will be included in the phase I part of this clinical trial.

Additional patients will be included in the expansion cohort up to a total of 15 patients. The expansion cohort will serve to further evaluate safety simultaneously with preliminary efficacy.

Patients will be selected and included in the study after testing the response to the drug with the Vivia Biotech ex vivo CDx PharmaFlow PM test. PharmaFlow PM test is a companion diagnostic (CDx) tool that provides a complete pharmacological profile for each individual, allowing the detection of patients resistant to OPB-111077 and enriching the study in patients that respond to the drug. The third of patients more sensitive to OPB-11077 wil be included in the study.

DETAILED DESCRIPTION:
The optimal management of relapsed AML in patients who are not candidates for HSCT has yet to be delineated. Given the median age at which AML is diagnosed and the high incidence of relapse and significant toxicities associated with standard intensive remission induction chemotherapy, new treatment options are needed to optimize AML outcomes. Changes on metabolism are critical in Acute Myeloid Leukaemia (AML); besides, leukemic cells have high requirements of energy and high basal metabolism. For this reason we hypothesized that deregulations of energy metabolism and mitochondria could play a central role in AML. OPB-111077, a novel low-molecular-weight compound discovered by Otsuka Pharmaceutical Co, Ltd, is a new class drug targeting cancer cell metabolisms and STAT3 and is being developed as an orally active antitumor agent for the treatment of various cancers. Sufficient preclinical studies have shown its activity in several types of tumors and especially in AML. Although in a phase I study their activity has been small in a group solid tumor, we may hypostatize that this drug could be more efficient in tumor cells with a high proliferative index as AML.

This is an open-label, phase Ib dose-escalation clinical trial to evaluate the safety and tolerability of oral OPB-111077 in AML relapsed or refractory to chemotherapy patients. OPB-111077 will be administered orally on a once daily dose schedule.

This open-label, nonrandomized trial will comprise 2 stages. A dose escalation stage will characterize the safety, tolerability and MTD, of OPB-111077. Subsequently, an expansion stage will further evaluate the safety and antitumor activity of OPB-111077 in AML relapsed or refractory to chemotherapy. The overall response rate of OPB-11077 in acute myeloid leukemia and its correlation with the ex-vivo PharmaFlow PM test will be also assessed.

Enrollment to the expansion cohort will begin following determination of the MTD.

OPB-111077 recommended dose for expansion cohort will be defined during the phase I as MTD. Intra patient dose escalation is not allowed at any time of the study.

Patients will be included in the study upon signed informed consent and will follow study procedures.

Two dose schemas will be employed:

* Level 1: 200 mg daily
* Level 2: 250 mg daily The starting dose level of oral OPB-111077 will be 200 mg od. A 3 + 3 dose-escalation scheme will be used.

A minimum of 3 patients will be initially enrolled per cohort. DLTs will be assessed during the DLT assessment window of 28 days following the first dose of OPB-111077. Patients who withdraw or are withdrawn from the study prior to completing the DLT assessment window for reasons other than a DLT will not be considered evaluable for DLT and will be replaced.

DLTs will be assessed during the DLT assessment window of 28 days following the first dose of OPB-111077. Patients who withdraw or are withdrawn from the study prior to completing the DLT assessment window for reasons other than a DLT will not be considered evaluable for DLT and will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old.
* Patients diagnosed of non M3 acute myeloid leukemia in relapse after intensive chemotherapy.
* Patients with a highest sensitivity (higher 70% of the samples analyzed) in the bone marrow analysis of the OPB-111077 ex-vivo sensitivity test.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Bilirubin ≤ 2 × Upper Limit of Normal (ULN). For subjects with known Gilbert's disease, bilirubin ≤ 3.0 mg/dL.
* Serum creatinine ≤2 × ULN or creatinine clearance (CrCl) ≥ 40 mL/min.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN.
* Left Ventricular Ejection Fraction (LVEF) must be equal to or greater than 50%.
* New York Heart Association (NYHA) congestive heart failure (CHF) class II or better.
* Recovery from adverse effects of prior therapy at time of enrollment to ≤ Grade 1 (excluding alopecia).
* Life expectancy ≥3 months
* Patients, or appropriate designee, must be able to provide informed consent.

Exclusion Criteria:

* Individuals with a history of other malignancies.
* Subject has uncontrolled intercurrent illness that would limit compliance with study requirements.
* Patients diagnosed of M3/Acute promyelocytic leukemia (APL).
* The subject has received systemic antineoplastic therapy within 14 days of study treatment.
* The subject has received any investigational agent within 28 days before the first dose of study treatment.
* The subject has not recovered to baseline or CTCAE ≤ Grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant Adverse Events (AEs).
* The subject has concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment.
* Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation.
* Malabsorption syndrome.
* Subject is unable to swallow capsules or tablets.
* Subject is pregnant or breastfeeding.
* Patients with history of allergic reactions attributed to components of OPB- 111077 that are not easily managed
* Subject has systemic infection requiring IV antibiotic therapy within 7 days preceding the first dose of study drug, or other severe infection.
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) of OPB-111077 in patients with in acute myeloid Leukemia. | 28 days
  Any adverse event related to the study drug that occurred during the first cycle and considered relevant:
  * Any Grade 3 or 4 non-hematologic toxicity
  * Any unexpected non-tolerable grade II adverse event possibly related to the treatment regimen that requires delay beyond 1 week until recovery
  * Hematological toxicity is not considered doses limiting due to the characteristic of Acute Myeloid Leukemia.

SECONDARY OUTCOMES:
Overall response rate. | Up to 8 months
  Percentage of patients to reach complete remission (CR), morphologic complete remission with incomplete blood count recovery (Cri) or partial remission (PR) according to Cheson et al criteria.
Overall response rate according to IC50 | Up to 8 months
  Percentage of patients to reach overall response rate according to IC50.
Overall response rate according to Area under de Curve | Up to 8 months
  Percentage of patients to reach overall response rate according to area under the curve.
Incidence of Treatment-Emergent Adverse Events | Up to 8 months
  Number of events per patient according to NCI CTCAE vs 4.03
Progression Free Survival | Up to 8 months
  Time from the date of informed consent form to the date of progression or death (from any cause), whichever occurs first
Overall Survival | Up to 12 months
  Time from the date of informed consent form to the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Martínez López, MD, Principal Investigator — Hospital 12 Octubre
Locations (6):
- Spain (6):
  - Hospital San Pedro Alcántara, Cáceres, Extremadura
  - MD Anderson Cancer Center, Madrid
  - Hospital 12 Octubre, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitario La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No